CLINICAL TRIAL: NCT04919317
Title: Enhanced Pain Control After Reduction Mammaplasty With Bupivicaine and Dexamethasone Regional Block: a Double-blind Randomized Controlled Trial
Brief Title: Combination Dexamethasone and Bupivacaine Pain Control in Reduction Mammaplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24361
Record Dates: First submitted 2021-05-21; First posted 2021-06-09 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Pain, Postoperative; Mammaplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial. Subjects were randomized 1:1 to the experimental or control groups. Each patient received the same Pecs II perineural block preoperatively with the same volume injected. Experimental group patients received 29mL 0.5% bupivacaine with 1mL of 4mg/mL dexamethasone, while control group patients received 29mL 0.5% bupivacaine with 1mL of 0.9% saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The surgeon (investigator), patient, and anesthesiologists were not aware of which arm each participant was assigned to. Furthermore, each injected analgesic was premixed and uniformly labeled to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator): Control group patients received 29mL bupivacaine plus 1mL 0.9% saline. Like the experimental group, 20mL of the mixture was injected into the fascial plane between the pectoralis minor and the serratus anterior muscles at the level of the third rib, while the remaining 10mL of the mixture was then injected into the fascial plane between the pectoralis major and pectoralis minor muscles during the same needlestick.
  Interventions: Drug: Saline
- Experimental (Experimental): Experimental group patients received 29mL bupivacaine plus 1mL of 4mg/mL dexamethasone. Like the control group, 20mL of the mixture was injected into the fascial plane between the pectoralis minor and the serratus anterior muscles at the level of the third rib, while the remaining 10mL of the mixture was then injected into the fascial plane between the pectoralis major and pectoralis minor muscles during the same needlestick.
  Interventions: Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: Dexamethasone 4mg — The experimental group received 4mg dexamethasone added to their bupivacaine block preoperatively just prior to bilateral reduction mammaplasty.
  Arms: Experimental
Drug: Saline — The control group received 1mL of 0.9% saline added to their bupivacaine block preoperatively just prior to bilateral reduction mammaplasty.
  Arms: Control

SUMMARY:
The addition of dexamethasone to non-liposomal bupivacaine in perineural blocks has been shown to enhance pain control and prolong the time until first request for postoperative narcotics in the fields of orthopedic, thoracic, and gynecologic surgery. This has not been investigated in any types of breast surgery. The investigators assessed if the combination of dexamethasone to bupivacaine in the preoperative field block prior to bilateral breast reduction surgery resulted in improved pain control relative to bupivacaine alone.

DETAILED DESCRIPTION:
The investigators conducted a double-blind randomized controlled trial to determine whether the addition of dexamethasone to bupivacaine in a preoperative Pecs II block resulted in improved pain control, relative to bupivacaine alone, in patients undergoing bilateral reduction mammaplasty.

Using a preassigned randomization list, patients were randomized to experimental and control groups in a ratio of 1:1 upon enrollment. Both groups received PECS II bupivacaine field blocks in the preoperative holding area, performed by an acute pain fellowship-trained anesthesiologist. The experimental group received 29mL of 0.5% bupivacaine mixed with 1mL 4mg/mL dexamethasone per side. The control group received 29mL 0.5% bupivacaine mixed with 1mL 0.9 saline solution per side. To maintain the blinded aspect of the study, the anesthesiologists were given pre-mixed vials labelled uniformly for the trial, regardless of the patient's treatment arm.

The patients all underwent bilateral breast reduction with a single surgeon. Postoperative pain regimens were standardized. Subjective pain scores, narcotic consumption, 4-hour interval vital signs, anti-emetic usage, and postoperative quality of life via an sf-36 questionnaire were all recorded per patient.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-80
* Bilateral reduction mammaplasty
* American Society of Anesthesiologists (ASA) physical status classification 1, 2, or 3
* Must choose to receive preoperative nerve block as part of pain management strategy

Exclusion Criteria:

* Allergy to dexamethasone or bupivacaine
* History of postoperative nausea and vomiting following anesthesia
* History of chronic pain conditions
* History of narcotic abuse or dependency
* History of chronic renal disease
* History of chronic liver disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Gassman, MD, FACS, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to other researchers if necessary
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after any potential publications from this study

REFERENCES:
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Broyles JM, Tuffaha SH, Williams EH, Glickman L, George TA, Lee Dellon A. Pain after breast surgery: Etiology, diagnosis, and definitive management. Microsurgery. 2016 Oct;36(7):535-538. doi: 10.1002/micr.30055. Epub 2016 Apr 4. PMID 27043853
- [Background] Ahiskalioglu A, Yayik AM, Demir U, Ahiskalioglu EO, Celik EC, Ekinci M, Celik M, Cinal H, Tan O, Aydin ME. Preemptive Analgesic Efficacy of the Ultrasound-Guided Bilateral Superficial Serratus Plane Block on Postoperative Pain in Breast Reduction Surgery: A Prospective Randomized Controlled Study. Aesthetic Plast Surg. 2020 Feb;44(1):37-44. doi: 10.1007/s00266-019-01542-y. Epub 2019 Nov 18. PMID 31741068
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Vetriselvan P, Mandal B, Bhatia N, Jain V. Effect of dexamethasone on analgesic efficacy of transverse abdominis plane block in laparoscopic gynecological procedures: A prospective randomized clinical study. J Anaesthesiol Clin Pharmacol. 2019 Apr-Jun;35(2):165-169. doi: 10.4103/joacp.JOACP_374_17. PMID 31303703
- [Background] Maher DP, Serna-Gallegos D, Mardirosian R, Thomas OJ, Zhang X, McKenna R, Yumul R, Zhang V. The Combination of IV and Perineural Dexamethasone Prolongs the Analgesic Duration of Intercostal Nerve Blocks Compared with IV Dexamethasone Alone. Pain Med. 2017 Jun 1;18(6):1152-1160. doi: 10.1093/pm/pnw149. PMID 27473629
- [Background] Bjorn S, Linde F, Nielsen KK, Borglum J, Hauritz RW, Bendtsen TF. Effect of Perineural Dexamethasone on the Duration of Single Injection Saphenous Nerve Block for Analgesia After Major Ankle Surgery: A Randomized, Controlled Study. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):210-216. doi: 10.1097/AAP.0000000000000538. PMID 28033159
- [Background] Ibrahim AS, Aly MG, Farrag WS, Gad El-Rab NA, Said HG, Saad AH. Ultrasound-guided adductor canal block after arthroscopic anterior cruciate ligament reconstruction: Effect of adding dexamethasone to bupivacaine, a randomized controlled trial. Eur J Pain. 2019 Jan;23(1):135-141. doi: 10.1002/ejp.1292. Epub 2018 Aug 6. PMID 30066465

RESULTS

PARTICIPANT FLOW:
Period: Hospitalization and Wound Follow-up
Arm/Group | Control | Experimental
Started | 26 | 30
Completed | 26 | 25 (5 patients completed the study but should not have been enrolled as they met pre-study exclusion criteria (chronic pain due to fibromyalgia))
Not Completed | 0 | 5
Not completed — Protocol Violation | 0 | 5
Period: SF-36 Quality of Life Survey Completion
Arm/Group | Control | Experimental
Started | 26 | 25
Completed | 14 | 19
Not Completed | 12 | 6
Not completed — Lost to Follow-up | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.73 (13.44) | 42.48 (15.17) | 40.57 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 7 | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.65 (10.12) | 34.12 (13.99) | 33.37 (12.07)
Anemia [Count of Participants; unit: Participants] | 4 | 5 | 9
Anxiety [Count of Participants; unit: Participants] | 4 | 5 | 9
Asthma [Count of Participants; unit: Participants] | 4 | 7 | 11
Depression [Count of Participants; unit: Participants] | 5 | 3 | 8
Degenerative Disc Disease [Count of Participants; unit: Participants] | 1 | 1 | 2
Degenerative Joint Disease [Count of Participants; unit: Participants] | 0 | 2 | 2
Diabetes [Count of Participants; unit: Participants] | 3 | 2 | 5
Drug Abuse [Count of Participants; unit: Participants] | 0 | 1 | 1
Gastroesophaageal reflux disease (GERD) [Count of Participants; unit: Participants] | 1 | 4 | 5
Hypothyroidism [Count of Participants; unit: Participants] | 0 | 3 | 3
Hyperlipidemia [Count of Participants; unit: Participants] | 1 | 4 | 5
Human immunodeficiency virus infection (HIV) / Acquired immunodeficiency syndrome AIDS [Count of Participants; unit: Participants] | 0 | 1 | 1
Hypertension [Count of Participants; unit: Participants] | 3 | 6 | 9
Insomnia [Count of Participants; unit: Participants] | 1 | 1 | 2
Migraines [Count of Participants; unit: Participants] | 1 | 5 | 6
Polycystic ovaries [Count of Participants; unit: Participants] | 0 | 1 | 1
Uterine Fibroids [Count of Participants; unit: Participants] | 0 | 1 | 1
Abnormal Uterine Bleeding [Count of Participants; unit: Participants] | 0 | 1 | 1
Rheumatoid Arthritis [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Initial Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded immediately upon arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 25
score on a scale | 8.3 (1.5) | 7.4 (2.1)

2. Primary Outcome: 4-hour Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded at 4-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 25
score on a scale | 5.5 (3.5) | 4.6 (3.6)

3. Primary Outcome: 8-hour Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded at 8-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 25
score on a scale | 4.4 (3.9) | 3.5 (3.6)

4. Primary Outcome: 12-hour Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded at 12-hours after arrival to the post-anesthesia recovery unit (PACU)
Population: Between the prior time point and this time point, 8 patients from the experimental group had been discharged to home
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 17
score on a scale | 3.9 (3.7) | 3.4 (3.6)

5. Primary Outcome: 16-hour Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded at 16-hours after arrival to the post-anesthesia recovery unit (PACU)
Population: Between the prior time point and this time point, 9 patients in the control group and 2 patients from the experimental group had been discharged to home
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 17 | 15
score on a scale | 5.6 (2.8) | 5.4 (2.8)

6. Primary Outcome: 20-hour Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded at 20-hours after arrival to the post-anesthesia recovery unit (PACU)
Population: Between the prior time point and this time point, 7 patients in the control group and 4 patients from the experimental group had been discharged to home
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 10 | 11
score on a scale | 5.8 (3.4) | 4.9 (3.8)

7. Primary Outcome: 24-hour Visual Analog Scale (VAS) Pain Scores
Description: Patient-reported pain scores on a scale of 1-10 (1 is low or no pain and 10 is the highest amount of pain)
Time Frame: Recorded at 24-hours after arrival to the post-anesthesia recovery unit (PACU)
Population: Between the prior time point and this time point, 4 patients in the control group and 6 patients from the experimental group had been discharged to home
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 6 | 5
score on a scale | 5.2 (3.8) | 8 (1.4)

8. Primary Outcome: Narcotic Consumption
Description: Mean narcotics used by each patient while in the hospital during the 24-hour hospitalization
Time Frame: Up to 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalents (OME)
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 25
Oral Morphine Equivalents (OME) | 36.60 (23.99) | 23.19 (17.26)

9. Secondary Outcome: Initial Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded immediately upon arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 24 | 25
mmHg | 124.2 (14.8) | 123.8 (13.5)

10. Secondary Outcome: 4-hour Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded at 4-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 18 | 19
mmHg | 118.0 (10.8) | 119.6 (16.4)

11. Secondary Outcome: 8-hour Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded at 8-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 20 | 19
mmHg | 113.8 (12.2) | 117.9 (17.4)

12. Secondary Outcome: 12-hour Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded at 12-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 18 | 23
mmHg | 106.7 (8.6) | 112.0 (17.8)

13. Secondary Outcome: 16-hour Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded at 16-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 16 | 19
mmHg | 112.3 (13.6) | 104.2 (8.0)

14. Secondary Outcome: 20-hour Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded at 20-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 13 | 15
mmHg | 106.5 (12.5) | 114.7 (9.6)

15. Secondary Outcome: 24-hour Blood Pressure
Description: Systolic blood pressure
Time Frame: Recorded at 24-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Experimental
Number analyzed (Participants) | 3 | 3
mmHg | 108.7 (8.5) | 118.3 (24.5)

16. Secondary Outcome: Initial Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded immediately upon arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 23 | 23
percentage of blood oxygen saturation | 99.4 (1.1) | 98.6 (2.1)

17. Secondary Outcome: 4-hour Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded at 4-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 18 | 19
percentage of blood oxygen saturation | 97.8 (1.6) | 96.9 (1.7)

18. Secondary Outcome: 8-hour Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded at 8-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 20 | 19
percentage of blood oxygen saturation | 98.7 (1.4) | 96.5 (2.0)

19. Secondary Outcome: 12-hour Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded at 12-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 18 | 23
percentage of blood oxygen saturation | 97.8 (1.5) | 97.0 (2.1)

20. Secondary Outcome: 16-hour Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded at 16-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 16 | 19
percentage of blood oxygen saturation | 98.8 (1.2) | 96.9 (1.6)

21. Secondary Outcome: 20-hour Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded at 20-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 12 | 13
percentage of blood oxygen saturation | 99.0 (0.9) | 98.3 (1.9)

22. Secondary Outcome: 24-hour Oxygen Saturation
Description: SpO2 as measured by pulse oximetry
Time Frame: Recorded at 24-hours after arrival to the post-anesthesia recovery unit (PACU)
Measure: Mean (Standard Deviation); unit: percentage of blood oxygen saturation
Arm/Group | Control | Experimental
Number analyzed (Participants) | 3 | 3
percentage of blood oxygen saturation | 99.3 (0.6) | 97.3 (3.1)

23. Secondary Outcome: Number of Patients Administered Anti-emetics at 4-hour Intervals
Description: Frequency of anti-emetics administered for complaints of nausea or vomiting at 4-hour intervals
Time Frame: Initial, 4, 8, 12, 16, 20, and 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 25
Participants
  Initial | 4 | 5
  4-hours postoperatively | 7 | 2
  8-hours postoperatively | 2 | 1
  12-hours postoperatively | 4 | 0
  16-hours postoperatively | 0 | 0
  20-hours postoperatively | 0 | 0
  24-hours postoperatively | 0 | 0

24. Secondary Outcome: Short-form 36-item (Sf-36) Quality of Life Questionnaire
Description: Aggregate results of the sf-36 quality of life assessment. This was provided one time to each patient, as early as at the first postoperative visit or at any time thereafter up to 2 months postoperatively. This assessment has been validated to measure 8 categories related to quality of life: physical functioning, limitations due to physical health, limitations due to emotional health, perceived level of energy/fatigue, emotional well-being, social functioning, pain, and overall general health. The responses to the 36 questions are tabulated and each category is given a score from 1-100 for each individual patient. Higher scores indicate a better quality of life for that category. The rows/data below report the mean and standard deviations of the collected scores in each category.
Time Frame: 1 week to 2 months postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 14 | 19
score on a scale
  Physical Functioning | 88.93 (15.83) | 90.42 (13.98)
  Limitations Due to Physical Health | 82.14 (24.86) | 79.17 (32.61)
  Limitations Due to Emotional Health | 88.10 (28.06) | 80.56 (32.04)
  Energy/Fatigue | 54.64 (12.63) | 52.92 (16.61)
  Emotional Well-being | 65.71 (6.41) | 59.00 (13.16)
  Social Functioning | 92.50 (9.71) | 88.75 (16.70)
  Pain | 59.64 (35.84) | 64.42 (25.16)
  Overall General Health | 51.43 (13.36) | 56.25 (13.69)

25. Secondary Outcome: Rate of Wound Complications
Description: Assessment of wound complications during any postoperative clinic visit
Time Frame: 1 week to 2 months postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 26 | 25
Participants
  None | 19 | 19
  Minor | 5 | 3
  Moderate | 2 | 2
  Severe | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 months postoperatively
Description: Other adverse event: wound complications of any severity
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 7/26 | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=26) | Experimental (N=25)
Wound complications (Surgical and medical procedures) | 7 | 8 — Assessment of wound complications during any postoperative clinic visit

LIMITATIONS AND CAVEATS:
Single-center study, which may limit the generalizability of the results The patient population is predominantly composed of racial minority communities, which may also limit the generalizability to many institutions Low SF-36 completion limited an adequate determination of the effects of the block on quality of life metrics. Some SF-36 questionnaires were completed by phone interview The COVID-19 pandemic halted enrollment for four months, which may have imposed a selection bias

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04919317/Prot_SAP_000.pdf